CLINICAL TRIAL: NCT07045519
Title: The Acute Effects of Local Vibration Application to the Gastrocnemius Muscle on Gait and Balance in Individuals With Hemiparetic Cerebral Palsy
Brief Title: Vibration Effects on Gait and Balance in CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Saniye Aydoğan Arslan, Kırıkkale University, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KırıkkaleBetulYılmaz; Betül Şevval Yılmaz (Other: Kırıkkale Üniversitesi)
Record Dates: First submitted 2025-05-16; First posted 2025-07-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy Hemiparetic Cerebral Palsy Spasticity Gait Disorders, Neurologic Postural Balance Impairment
Keywords: Hemiparetic Cerebral Palsy; Randomized Controlled Trial; Modified Ashworth Scale; Tardieu Scale; Gross Motor Function; Pediatric Physiotherapy; Gait Analysis; Balance Assessment; Gastrocnemius Muscle; Spasticity; Local Vibration Therapy
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Local Vibration Therapy (Experimental): Participants in the treatment group will receive local vibration applied for 10 minutes to the most prominent area of the spastic medial gastrocnemius muscle.
  Interventions: Device: Local Vibration Therapy
- Placebo Comparator: Sham Vibration (Placebo Comparator): Participants in the placebo group will be placed in the prone position and the vibration device will be placed on the same area as in the treatment group for 10 minutes without delivering any vibration.
  Interventions: Device: Sham Vibration

INTERVENTIONS:
Device: Local Vibration Therapy — Local vibration (LV) will be applied using the Vibrasens© device (Techno Concept, Mane, France). Vibrasens© is a non-invasive therapeutic mechanical vibrator used for transcutaneous vibratory stimulation in sensorimotor rehabilitation. The system includes one pilot unit, one manual vibrator (VB200), four flat skin contactors for tendon applications, four round skin contactors for surface applications, a power supply, a user manual, and a protocol guide.
  Arms: Experimental: Local Vibration Therapy
Device: Sham Vibration — Participants will receive sham stimulation by placing the Vibrasens© device on the same area as the treatment group for 10 minutes, without activating the vibration function. They will be informed that they will only feel the contact of the device.
  Arms: Placebo Comparator: Sham Vibration

SUMMARY:
This randomized controlled study aims to investigate the acute effects of local vibration applied to the spastic medial gastrocnemius muscle on balance and spatiotemporal gait parameters in children with hemiparetic cerebral palsy. Children aged 4 to 18 years with spasticity levels of 1 to 2 on the Modified Ashworth Scale and Gross Motor Function Classification System (GMFCS) levels I-II will be included. Participants will be randomly assigned to either a treatment group receiving local vibration or a placebo group. Assessments will be conducted before, immediately after, and 30 minutes after the intervention. Balance will be assessed using the Timed Up and Go Test (TUG), Pediatric Reach Test, Tandem Stance Test, and Pediatric Berg Balance Scale. Spatiotemporal gait parameters will be measured using a digital gait analysis system. The results will provide insights into the immediate effectiveness of localized vibration therapy in pediatric cerebral palsy rehabilitation.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) are known to have postural control deficits and motor impairments, primarily due to damage in brain areas responsible for postural regulation. These deficits often lead to balance and orientation problems, particularly affecting motor tasks such as walking. Despite various therapeutic approaches, many children with CP continue to experience difficulties in achieving independent ambulation.

Recent studies have shown that vibration therapy may enhance walking performance in children with CP. Local vibration applied to the spastic gastrocnemius muscle has been associated with improvements in muscle tone, functional gait parameters, and electromyographic patterns. However, the literature is predominantly focused on whole-body vibration and its effects on spasticity. There is a lack of research specifically examining the effects of local vibration on balance and gait parameters in individuals with spastic CP.

This randomized controlled trial aims to investigate the acute effects of local vibration applied to the spastic gastrocnemius muscle on balance and spatiotemporal gait parameters in children with hemiparetic cerebral palsy.

Participants will be recruited from a private special education and rehabilitation center. Sample size will be determined based on a power analysis following a pilot study. Individuals classified as Level I or II according to the Gross Motor Function Classification System (GMFCS) will be included. Participants will be randomly assigned to either the treatment or placebo group using a coin-flip method. Evaluations will be conducted before the intervention, immediately after, and 30 minutes post-intervention.

Demographic and clinical information such as age, gender, type of CP, use of assistive devices, history of surgery, and orthopedic deformities will be recorded. Assessments will be performed by experienced physiotherapists.

Balance will be assessed using the Timed Up and Go Test (TUG), Pediatric Reach Test, and Tandem Stance Test. Spatiotemporal gait parameters will be analyzed using a wireless miniature digital gait analysis system.

Inclusion Criteria:

* Children aged 4-18 years diagnosed with hemiparetic CP,
* GMFCS Level I-II (ambulatory without support),
* Spasticity in the gastrocnemius muscle (Modified Ashworth Scale 1, 1+, or 2),
* Able to follow verbal instructions,
* No Botox treatment in the last 3 months or surgery in the last 6 months,
* Voluntary participation with informed parental consent.

Exclusion Criteria:

* Botox treatment or surgery for spasticity within the past 6 months,
* Neurological disorders other than CP, joint pain, or fracture history affecting independent standing/walking,
* Severe intellectual disability preventing compliance,
* Behavioral problems during assessment,
* Lack of consent.

Assessment Parameters:

* Balance: Pediatric Berg Balance Scale (PBBS), Timed Up and Go Test (TUG), Pediatric Reach Test, Tandem Stance, Single-leg Stance.
* Gross Motor Function: Gross Motor Function Measure (GMFM).
* Spasticity: Modified Ashworth Scale (MAS), Modified Tardieu Scale (MTS).
* Gait Analysis: Spatiotemporal parameters via digital gait analysis system.

The Modified Tardieu Scale will be used to measure the quality and angle of muscle reaction to passive stretch at three different velocities (V1, V2, V3).

The Pediatric Berg Balance Scale consists of 14 items scored from 0 to 4, evaluating functional balance in daily life activities.

The digital gait analysis system uses an accelerometer-based sensor attached to the pelvis to measure walking parameters.

Intervention Protocol:

Treatment Group:

Local vibration will be applied to the most prominent area of the spastic medial gastrocnemius muscle using the Vibrasens® (Techno Concept, France). The device delivers non-invasive mechanical vibrations. A 10-minute session of local vibration at 80 Hz with 1 mm amplitude will be administered.

Placebo Group:

The device will be placed on the same muscle area for 10 minutes without delivering vibration. Participants will only feel the contact of the device.

Statistical Analysis:

* Continuous variables will be expressed as mean ± standard deviation.
* Shapiro-Wilk test will assess normality.
* Independent t-test or Mann-Whitney U test will compare groups depending on data distribution.
* Chi-square test will be used for categorical variables.
* Within-group comparisons will use paired t-tests or Wilcoxon tests as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy, classified as GMFCS Level I or II
* Aged between 4 and 18 years
* Presence of spasticity in the gastrocnemius muscle (Modified Ashworth Scale score of 1, 1+, or 2)
* Able to walk independently
* Ability to follow verbal instructions
* No botulinum toxin injection in the past 3 months
* No lower limb surgery in the past 6 months
* Voluntary participation with written and verbal informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Botulinum toxin injection or surgical intervention for spasticity within the past 6 months
* Neurological disorders other than cerebral palsy
* Musculoskeletal problems that may affect standing or walking (e.g., joint pain, lower extremity fractures within the past 6 months)
* Severe cognitive impairment preventing understanding of basic commands
* Behavioral problems or poor cooperation that interfere with assessments
* Lack of written informed consent from parents or legal guardians

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Modified Tardieu Scale (MTS) | Baseline and immediately after intervention
  The MTS is a clinical tool used to assess spasticity. Although not as commonly used as the Modified Ashworth Scale (MAS), it is considered a more effective method for evaluating spasticity because it measures resistance to passive movement at two different velocities (Tardieu et al., 1999).
  The Modified Tardieu Scale includes:
  Quality of muscle reaction (X): Rated on a scale from 0 (no resistance to passive movement) to 5 (joint is immobile).
  Angle of muscle reaction (Y): Measured with a goniometer relative to the position in which the muscle is at its shortest length.
  Stretching velocities: The assessment is performed at three different velocities: V1 (slow), V2 (gravity), and V3 (fast) (Tardieu et al., 1999; Patrick & Ada, 2006).
Gross Motor Function Classification System (GMFCS): | Baseline
  The GMFCS evaluates sitting, transfers, and mobility. It classifies children based on their age and motor skills. The system includes five levels that clearly define functional differences (Palisano et al., 2008).
  The Turkish version of the GMFCS was developed by Kerem Günel and colleagues.
  Levels:
  Level I: Walks without limitations.
  Level II: Walks with limitations.
  Level III: Walks using a hand-held mobility device.
  Level IV: Self-mobility is limited; may use powered mobility.
  Level V: Transported in a manual wheelchair (Günel et al., 2010).
Pediatric Berg Balance Scale (PBBS): | Baseline
  The PBBS is a modified version of the original Berg Balance Scale, adapted by Franjoine et al. for use in children. It is used to evaluate functional balance during daily living activities (Franjoine et al., 2003).
  The PBBS consists of 14 items, each scored from 0 to 4. The Turkish version was published by Erden et al. (2011).
Timed Up and Go Test (TUG): | Baseline and immediately after intervention
  The TUG test assesses postural control, walking speed, functional mobility, and balance in children with cerebral palsy (Rose et al., 2011). During the test, the child rises from a chair, walks 10 meters, turns around, and returns to sit down. The test is timed with a stopwatch.
10-Meter Walk Test (10MWT): | Baseline and immediately after intervention
  This test measures the time it takes for an individual to walk 10 meters at a self-selected comfortable pace. It is commonly used to guide rehabilitation planning in individuals with cerebral palsy (Li et al., 2012).
Pediatric Reach Test | Baseline and immediately after intervention
  This test evaluates the dynamic component of balance. Children are asked to reach forward and sideways without lifting their heels, and the distance is measured in centimeters (Fay et al., 2007).
Tandem Stance Test | Baseline and immediately after intervention
  The child is instructed to stand with one foot placed heel-to-toe in front of the other. The test is conducted in two phases: with eyes open and with eyes closed (Franjoine et al., 2003).

SECONDARY OUTCOMES:
Walking Speed (m/s) | Baseline and immediately after intervention
  Walking speed will be measured using a digital gait analysis system equipped with a pelvic accelerometer to assess functional mobility.
Step Length (cm) | Baseline and immediately after intervention
  Step length, defined as the distance between successive footfalls of alternate feet, will be measured using the digital gait analysis system.
Stride Length (cm) | Baseline and immediately after intervention
  Stride length, the distance between successive footfalls of the same foot, will be assessed using a pelvic accelerometer during gait analysis.
Cadence (steps/min) | Baseline and immediately after intervention
  Cadence will be measured as the number of steps taken per minute during a walking trial using a digital gait analysis system.
Double Support Time (s) | Baseline and immediately after intervention
  Double support time, defined as the duration both feet are in contact with the ground during walking, will be measured using gait analysis.
Stance Time (s) | Baseline and immediately after intervention
  Stance time, the duration one foot remains in contact with the ground during a gait cycle, will be assessed to determine temporal gait stability.
Swing Time (s) | Baseline and immediately after intervention
  Swing time, defined as the period during which a foot is off the ground, will be measured for each leg using gait analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Yıldırım Beyazıt University, Ankara
  - Kırıkkale University, Kırıkkale